CLINICAL TRIAL: NCT07250997
Title: Study of the Effectiveness of the PALLAS Laser in the Treatment of Skin Diseases That Respond Well to UV Light
Brief Title: PALLAS Laser for Skin Diseases
Acronym: PALLAS-UV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Kemény Lajos, Professor, MD, DSc, MHAS, Szeged University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD-PALL-01; CIV-HU-25-08-053914 (Other: National Centre for Public Health and Pharmacy, Budapest)
Record Dates: First submitted 2025-09-23; First posted 2025-11-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Vitiligo Vulgaris; Psoriasis; Alopecia Areata; Atopic Dermatitis
Keywords: UVB laser treatment; PALLAS laser; vitiligo; psoriasis; alopecia areata; atopic dermatitis
MeSH Terms: conditions — Vitiligo; Psoriasis; Alopecia Areata; Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pallas Laser treated (Other): UVB treated patients
  Interventions: Device: UVB laser treatment

INTERVENTIONS:
Device: UVB laser treatment — In clinical practice, 311 nm ultraviolet B (UVB) phototherapy is often used to treat various skin conditions. In 1996, the 308 nm xenon chloride excimer laser was developed for the treatment of psoriasis. In the last decades, excimer treatment has been incorporated into international therapeutic protocols for the treatment of psoriasis alongside conventional 311 nm UVB therapies. In the present study, the investigators aim to gain experience with a UVB laser (Pallas) operating at a wavelength of 311 nm. The CE-marked Pallas UVB laser will be used for the same indications as the 308 nm excimer laser. The procedure is not new, but the significance of this study lies in its potential to provide us with experience using this device for targeted UVB treatment.

SUMMARY:
The primary objective of this study is to get clinical experiences with the PALLAS laser in the treatment of skin conditions that respond well to UV light (vitiligo, psoriasis, alopecia areata, atopic dermatitis).

The secondary objective is to assess how user-friendly is the Pallas laser in the treatment of skin diseases.

The patient in the trial will receive UVB laser treatment (2 treatments per week for up to 3 months). The treatments will be carried out by the doctors participating in the trial.

The treatment takes approximately 10 minutes per session, and can last up to 3 months per patient.

Photographic documentation of the lesions to be treated and the lesions treated is taken at the start of the examination and then once a month.

At the end of the study, the patient rates the treatment and improvement on a Patient Satisfaction Scale.

DETAILED DESCRIPTION:
This clinical study is a prospective testing and assessment of a CE marked PALLAS laser device within its intended use, carried out in one centre.

PALLAS is a solid-state ultraviolet laser system with 311 nm emission wavelength for tissue incision, destruction and removal.

The laser is intended for use on different parts of the skin, typically the face, hands, arms, feet or legs.

Pallas eliminates the shortcomings of currently used excimer lasers, such as the instability of the emitted energy and the expensive maintenance costs. The energy emitted by the laser is stable over a long period of time, maximising the effectiveness of the treatments and minimising the potential side effects of skin burns.

EUDAMED registration

LASEROPTEK sheet with SRN number:

https://ec.europa.eu/tools/eudamed/#/screen/search-eo/61c45e80-9297-4dcd-8940-8f7ccad5ef22 Actor ID/SRN: KR-MF-000018426

ELIGIBILITY:
Inclusion Criteria:

1. The subject understands the information provided, gives informed consent to participate in the study and is deemed by the investigator to be able to participate,
2. a skin condition that is expected to respond well to targeted UVB treatment,
3. a signed consent form.

Exclusion Criteria:

1. Patient under 18 years of age,
2. pregnancy
3. epilepsy,
4. fever, infectious diseases,
5. the patient is within one month or currently enrolled in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: visible improvement of the treated skin disease. | maximum 3 months
  Vitiligo (VES score): https://www.vitiligo-calculator.com/ Psoriasis (PASI-score): https://pasi.corti.li/ Alopecia areata (SALT score) https://dermatopics.dk/salt-score/ Atopiás dermatitis (EASI score): https://www.easiderm.com/

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | Maximum 3 months
  The Dermatology Life Quality Index (DLQI) is a 10-question, self-administered survey that assesses how skin diseases affect a patient's health-related quality of life.

OTHER OUTCOMES:
Patient Satisfaction Score | maximum 3 months
  At the last visit, the patient assesses the improvement:
  Patient satisfaction scale:
  0 = extremely dissatisfied
  1. = dissatisfied
  2. = satisfied
  3. = extremely satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Albert Szent-Györgyi Clinical Centre, Department of Dermatology and Allergology, Szeged, Csongrád-Csanád Vármegye, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baltas E, Csoma Z, Ignacz F, Dobozy A, Kemeny L. Treatment of vitiligo with the 308-nm xenon chloride excimer laser. Arch Dermatol. 2002 Dec;138(12):1619-20. No abstract available. PMID 12472364
- [Background] Bonis B, Kemeny L, Dobozy A, Bor Z, Szabo G, Ignacz F. 308 nm UVB excimer laser for psoriasis. Lancet. 1997 Nov 22;350(9090):1522. doi: 10.1016/S0140-6736(05)63945-1. No abstract available. PMID 9388408
- [Background] Baltas E, Nagy P, Bonis B, Novak Z, Ignacz F, Szabo G, Bor Z, Dobozy A, Kemeny L. Repigmentation of localized vitiligo with the xenon chloride laser. Br J Dermatol. 2001 Jun;144(6):1266-7. doi: 10.1046/j.1365-2133.2001.04248.x. No abstract available. PMID 11422057